CLINICAL TRIAL: NCT03483363
Title: Topical Antibiotic Irrigation (Gentamicin) in Prophylaxis of Midfacial Fracture Surgical Wounds
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment issues
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nagi Demian, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HSC-DB-18-0038
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Therapeutic Irrigation; Gentamicins; Saline Solution; Chemoprevention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- topical irrigation with the antibiotic plus intravenous (IV) prophylactic antibiotic (Experimental): Fractures will be topically irrigated with the topical antibiotic gentamicin (80mg diluted in 1L 0.9% normal saline) prior to closure.
  [previously, this arm involve topical irrigation with bacitracin topical antibiotic (50,000 units), but in April of 2020 the study was modified to use gentamycin rather than bacitracin, after the FDA warning of the toxic side effects of bacitracin and because the hospital where the study was conducted removed bacitracin from its formulary.]
  Interventions: Drug: topical irrigation with gentamicin (80mg diluted in 1L 0.9% normal saline); Drug: intravenous (IV) prophylactic antibiotic
- topical irrigation with sterile normal saline (NS) plus intravenous (IV) prophylactic antibiotic (Active Comparator): Fractures will be irrigated with sterile normal saline prior to closure. All groups with receive standard parenteral (IV) prophylactic antibiotic.
  Interventions: Drug: topical irrigation with sterile normal saline (NS); Drug: intravenous (IV) prophylactic antibiotic

INTERVENTIONS:
Drug: topical irrigation with gentamicin (80mg diluted in 1L 0.9% normal saline) — Fractures will be irrigated with the topical antibiotic gentamicin (80mg diluted in 1L 0.9% normal saline) prior to closure.
  Arms: topical irrigation with the antibiotic plus intravenous (IV) prophylactic antibiotic
Drug: topical irrigation with sterile normal saline (NS) — Fractures will be irrigated with sterile normal saline prior to closure.
  Arms: topical irrigation with sterile normal saline (NS) plus intravenous (IV) prophylactic antibiotic
Drug: intravenous (IV) prophylactic antibiotic — All arms with receive standard parenteral (IV) prophylactic antibiotic.

SUMMARY:
The purpose of this study is to evaluate the use of topical antibiotic irrigation (gentamycin) and its ability to reduce surgical site infections in midfacial fracture surgery compared to sterile normal saline (NS).

Previously, this study evaluated a different antibiotic, bacitracin, but in April of 2020 the study was modified to use gentamycin rather than bacitracin, after the FDA warning of the toxic side effects of bacitracin and because the hospital where the study was conducted removed bacitracin from its formulary.

ELIGIBILITY:
Inclusion Criteria:

* patients who are planned for open reduction internal fixation of midfacial fractures as part of standard of care
* patients who are admitted to Memorial Hermann hospital at Texas Medical Center
* able to sign their own consent

Exclusion Criteria:

* infected surgical sites
* allergies to bacitracin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Demian, MDDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Irrigation With the Antibiotic Plus Intravenous (IV) Prophylactic Antibiotic: Fractures will be topically irrigated with the topical antibiotic gentamicin (80mg diluted in 1L 0.9% normal saline) prior to closure.
  [previously, this arm involve topical irrigation with bacitracin topical antibiotic (50,000 units), but in April of 2020 the study was modified to use gentamycin rather than bacitracin, after the FDA warning of the toxic side effects of bacitracin and because the hospital where the study was conducted removed bacitracin from its formulary.]
  topical irrigation with gentamicin (80mg diluted in 1L 0.9% normal saline): Fractures will be irrigated with the topical antibiotic gentamicin (80mg diluted in 1L 0.9% normal saline) prior to closure.
  intravenous (IV) prophylactic antibiotic: All arms with receive standard parenteral (IV) prophylactic antibiotic.
Period: Overall Study
Arm/Group | Topical Irrigation With the Antibiotic Plus Intravenous (IV) Prophylactic Antibiotic | Topical Irrigation With Sterile Normal Saline (NS) Plus Intravenous (IV) Prophylactic Antibiotic
Started | 17 | 22
Completed | 17 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Irrigation With the Antibiotic Plus Intravenous (IV) Prophylactic Antibiotic | Topical Irrigation With Sterile Normal Saline (NS) Plus Intravenous (IV) Prophylactic Antibiotic | Total
Number analyzed (Participants) | 17 | 22 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.82 (15.06) | 37.81 (15.18) | 41.30 (15.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Infection (SSI)
Description: Surgical site infections include evidence of infection: persistent swelling, fever, recurrent swelling, erythema, and purulent discharge.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Irrigation With the Antibiotic Plus Intravenous (IV) Prophylactic Antibiotic | Topical Irrigation With Sterile Normal Saline (NS) Plus Intravenous (IV) Prophylactic Antibiotic
Number analyzed (Participants) | 17 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Topical Irrigation With the Antibiotic Plus Intravenous (IV) Prophylactic Antibiotic | Topical Irrigation With Sterile Normal Saline (NS) Plus Intravenous (IV) Prophylactic Antibiotic
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/22
Other Adverse Events (participants affected / at risk) | 0/17 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT03483363/Prot_SAP_000.pdf